CLINICAL TRIAL: NCT04100070
Title: Impact of an Intensive Monitoring on Glycaemic Control One Year After Initiating Continuous Subcutaneous Insulin Infusion in Children With Type 1 Diabetes.
Brief Title: Intensive Versus Standard One Year Monitoring on Glycaemic Control After Initiating CSII in Children With DT1. DEEP Study
Acronym: DEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ISIS Diabete Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A02932-53
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1; Pediatric ALL
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Prospective randomized parallel groups open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring (Other): Usual follow-up of children by pediatricians as recommended by relevant Authorities (HAS) both in terms of frequency of visits and rhythm of biological controls.
  Standard technical training, maintenance and monitoring by the CSII service provider as defined by the official specifications (LPPR)
  Interventions: Behavioral: Monitoring of the patients
- Intensive monitoring (Other): Usual follow-up of children by pediatricians as recommended by relevant Authorities (HAS) both in terms of frequency of visits and rhythm of biological controls completed by a personalized vision of the patient glycaemic data along the study.
  Intensive technical training, maintenance and monitoring by the CSII service provider with a higher frequency of contacts during the period (additional nurse visits).
  Interventions: Behavioral: Monitoring of the patients

INTERVENTIONS:
Behavioral: Monitoring of the patients — Follow-up of the patients during the 12 months study periods including :
  * visits with the diabetologist/pediatrician
  * contacts with the service provider (nurses' visits) (more in intensive group)
  * personalized monitoring of glycemic data transferred to the diabetologist/pediatrician for each visit (only in intensive group)

SUMMARY:
More than half of type 1 diabetes (DT1) children are under CSII (Continuous Subcutaneous Insulin Infusion).

Several studies showed that despite a patients' follow-up mostly by hospital-based paediatricians, there are still some concerns on long-term glycaemic control with inconstant results on glycaemic control either due to CSII adherence or nutrition management issues.

Consequently, this real life study aims to compare two monitoring methods (standard versus intensive) in children initiating a CSII treatment and assess the impact on glycaemic control after one year.

DETAILED DESCRIPTION:
As CSII becomes more and more the gold standard therapy in children with type 1 diabetes, there have been some questions regarding the long-term effect of these treatments with some concerns on the inconstant results on glycaemic control either due to CSII adherence or nutrition management issues.

The DCCT (Diabetes Control and Complications Trial) study has already shown in diabetic adults that intensification of treatment and follow-up could result in significative improvement of glycaemic control.

This study aims to test this hypothesis of significant improvement after one year following CSII initiation on glycaemic control.

Two parallel arms will be compared in real life conditions; one with standard recommendations-based follow-up by both diabetologists/pediatricians and service provider and the other with intensive follow-up with higher frequency of provider's nurses visits and personalization of patient status transferred to the physician for each diabetologists/pediatricians visit.

Thus, investigators could determine after one year if the glycaemic control is better with one or the other of these follow-up procedures.

Glycaemic control will be assessed both by the evolution of HbA1c during the study period and its last level at the end of the study. Its evaluation will be completed by counting of all symptomatic hypoglycemia occurence during the study.

ELIGIBILITY:
Inclusion Criteria:

* Children (<18 yo) with not controlled type 1 diabetes seen by diabetologists/paediatricians immediately following the initiation of CSII.
* Children for whom it is the first initiation of CSII.
* Children (or their parents if necessary) having read the information note and having dated and signed the informed consent form.

Exclusion Criteria:

* Children with a history of diabetes less than 12 months.
* Children with HbA1c values below 7.5 or above 10 before CSII initiation.
* Children treated by CSII for more than 3 months.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact on glycaemic control one year after CSII initiation | HbA1c values at inclusion and last known measurement at the 12 months last visit
  Evolution of HbA1c measurement between last measure before CSII initiation and 12 months after.
Impact on glycaemic control all along the study | Assessment and counting of all unplanned hospitalizations during the 12 months period
  Unplanned hospitalization rate during the study Severe hypoglycemia during the study period

SECONDARY OUTCOMES:
Impact on glycaemic control upon age classes | HbA1c values at inclusion and last known measurement at the 12 months last visit
  sub-groups based one age (<7 years old [yo], 7-12 yo, 13-17 yo)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Nicolino, MD PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Isis Diabete Service, Gennevilliers, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No